CLINICAL TRIAL: NCT00156416
Title: Menopause and Meditation for Breast Cancer Survivors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Susan Cohen, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21CA106336-01A1 (NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Menopause
Keywords: menopause; hot flash; night sweat; meditation; breast cancer
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation group (Experimental): Participants received 8 weeks of mindfulness meditation instruction and support
  Interventions: Behavioral: Mindfulness Meditation
- Education group (Active Comparator): Participants received 8 weeks of healthy living instruction
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Mindfulness Meditation — 8 weeks of meditation training

SUMMARY:
One of the consequences of breast cancer treatment for younger women is the abrupt onset of menopause and its related symptoms. Menopausal symptoms disrupt usual activities, alter sleep patterns and decrease quality of life. The purpose of this randomized feasibility pilot study is to examine mindfulness meditation for menopausal symptom management for women who are breast cancer survivors and for women with naturally occurring menopause. The study is designed to: 1. establish the feasibility of a mindfulness meditation program for women who experience menopausal symptoms (e.g. hot flushes). 2. explore the treatment benefit of a mindfulness meditation program for menopausal symptom relief using changes in frequency and severity of hot flushes; frequency of sleep disruption, various aspects of quality of life and physiologic stress response (cortisol) as outcome measures. 3. evaluate whether the treatment benefits of mindfulness meditation differ in menopausal women with naturally occurring menopause versus women with menopause secondary to chemotherapy for breast cancer. Participants randomized to the attention control group will be offered meditation training after completion of the intervention and follow up phases. Participants will attend 8 meditation sessions or 8 attention control sessions. Study variables are Menopausal Hot Flushes (self report & skin conductance monitoring), Sleep Disruption (Pgh Sleep Quality Index), Physiologic Stress Response (cortisol), Quality of Life (Menopausal Quality of Life); and Protocol Design (recruitment & retention rates, exit interviews). A convenience sample of 60 women who experience menopausal symptoms will be recruited.

DETAILED DESCRIPTION:
One of the consequences of breast cancer treatment for younger women is the abrupt onset of menopause and its related symptoms. Menopausal symptoms disrupt usual activities, alter sleep patterns and decrease quality of life. In light of the recent findings from the Women's Health Initiative (re:use of exogenous estrogen), the need to investigate non-hormonal approaches (meditation) for short-term menopausal symptom discomfort is high. The purpose of this randomized feasibility pilot study is to examine mindfulness meditation for menopausal symptom management for women who are breast cancer survivors and for women with naturally occurring menopause. The study is designed to: 1. establish the feasibility of a mindfulness meditation program for women who experience menopausal symptoms (e.g. hot flushes). 2. explore the treatment benefit of a mindfulness meditation program for menopausal symptom relief using changes in frequency and severity of hot flushes; frequency of sleep disruption, various aspects of quality of life and physiologic stress response (cortisol) as outcome measures. 3. evaluate whether the treatment benefits of mindfulness meditation differ in menopausal women with naturally occurring menopause versus women with menopause secondary to chemotherapy for breast cancer. A 2x2 factorial repeated design will be used. The four randomized groups will consist of 1) naturally occurring menopause meditation; 2) naturally occurring menopause attention control; 3) breast cancer survivors meditation; 4) breast cancer survivors attention. Participants randomized to the attention control group will be offered meditation training after completion of the intervention and follow up phases. Participants will attend 8 meditation sessions or 8 attention control sessions. Study variables are Menopausal Hot Flushes (self report & skin conductance monitoring), Sleep Disruption (Pgh Sleep Quality Index), Physiologic Stress Response (cortisol), Quality of Life (Menopausal Quality of Life); and Protocol Design (recruitment & retention rates, exit interviews). A convenience sample of 60 women who experience menopausal symptoms will be recruited. Data analysis includes descriptive statistics, repeated measures content analysis. Results from this feasibility pilot study will inform the design of a larger randomized clinical trial to test the effectiveness of mindfulness meditation as a self care intervention for menopausal symptom management and improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* . Subjects will be selected based on their self-identification of menopausal hot flushes. Subjects may identify other menopausal symptoms but must have hot flushes. Inclusion criteria will include English speaking, self-identification of the menopausal symptom of hot flushes following treatment for breast cancer (stage I or II) and amenorrhea secondary to breast cancer treatment or for women with naturally occurring menopause amenorrhea of greater that one year but less than three years.

Exclusion Criteria:

* Exclusion criteria are, for women with breast cancer, amenorrhea of greater that one year prior to their diagnosis of breast cancer. Also, excluded is concurrent treatment of menopausal symptoms with hormonal supplementation, herbal remedies, acupuncture, acupressure or non-hormonal pharmacologic agents prescribed at doses specifically for hot flush relief (beta blockers, SSRIs). However, women taking either serotonin reuptake inhibitors for depression or beta-blockers for hypertension who exhibit hot flushes sufficient to meet inclusion criteria will be accepted into the study. Previous treatment of menopausal symptoms with hormones, herbs or acupuncture, structured meditation and/or regular yoga practice must have ceased at least three months prior to enrollment in the study to allow for a sufficient wash out period. Women who are presently in chemotherapy treatment for breast cancer are excluded due to the potential confounding effect of mindfulness meditation on quality of life due to chemotherapy symptom relief. Women with a moderate to severe level of depression (>27), or suicidal thoughts or wishes, as measured by the Beck Depression Index, 2nd Ed (BDI-II), will be excluded and referred for treatment. However, following treatment for depression, they may enroll in the study assuming continuation of hot flushes at inclusion criteria levels.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
hot flushes | 21 weeks

SECONDARY OUTCOMES:
Sleep | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Cohen, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States